CLINICAL TRIAL: NCT02354924
Title: A Prospective Randomized Controlled Study to Evaluate the Clinical Performance of VISCO Soft Contact Lens on a Daily Wear Basis
Brief Title: Clinical Evaluation of Two Daily Wear Silicon Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visco Vision Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1000601M
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Visco soft contact lens (Experimental): Olifilcon A, Daily wear, monthly disposable soft contact lens
  Interventions: Device: Visco soft contact lens
- Biofinity soft contact lens (Active Comparator): Comfilcon A, Daily wear, monthly disposable soft contact lens
  Interventions: Device: Biofinity soft contact lens

INTERVENTIONS:
Device: Biofinity soft contact lens — Biofinity soft contact lens on two eyes and follow up for 3 months (90 days). It is necessary to remove contact lenses every day and replace after 30 days.
  Arms: Biofinity soft contact lens
Device: Visco soft contact lens — Viso soft contact lens on two eyes and follow up for 3 months (90 days). It is necessary to remove contact lenses every day and replace after 30 days.
  Arms: Visco soft contact lens

SUMMARY:
The purpose of this study is to demonstrate that the VISCO (Olifilcon A) soft contact lens could be prescribed as a supportive care for myopic persons.

DETAILED DESCRIPTION:
This randomized controlled study will involve at least 50 evaluable subjects divided evenly among 5 study sites in Taiwan. Each study site will enroll 12 subjects at least. The ration of evaluable test subjects to control subjects will be 2 to 1. Subjects who have normal ocular health and conform to a set of standard criteria will wear one of the study lenses on two eyes and follow up for 3 months (90 days). Lenses will be assigned to subject according to a predetermined randomized order. It is necessary to remove contact lenses every day and replace after 30 days. Any unscheduled visit will be allowed when there is a medication necessary. The data for slit lamp findings, symptoms/problems/complaints, keratometry (K) reading, refractive changes (absolute value), visual acuity data, average wear time (AWT), discontinuations, and lens replacement will be collected to claim that the VISCO Soft Contact Lens is as safe and effective as BIOFINITY (comfilcon A) Soft Contact Lens (CooperVision).

ELIGIBILITY:
Inclusion Criteria:

* Subject should have normal eyes and use no ocular medications
* Subject with -1.00 to -10.00 D myopia, less than -1.25 D astigmatism
* VA correctable to 20/25 or better.
* Willing to comply with all study procedures and be available for the duration of the study.
* Provide signed and dated informed consent form.

Exclusion Criteria:

* Subjects have history of allergies that would contraindicate solution use and/or "normal" contact lens wear.
* Cornea sensitivity low, high myopes, Keratoconus, dry eye with Schirmer Test < 5mm/5min or other physical condition that would contraindicate contact lens wear.
* Subjects have other active ocular or systemic disease that would contraindicate contact lens wear.
* Subjects have medications that would contraindicate contact lens wear.
* Females who are pregnant, breastfeeding, birth control pill taken or who intended to become pregnant over the course of the study.
* Current drug or alcohol use or dependence that would interfere with adherence to study requirements.
* Individuals participating in other clinical studies.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huey Chuan Cheng, MD. MS, Principal Investigator — Mackey Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Visco Soft Contact Lens: Olifilcon A, Daily wear, monthly disposable soft contact lens
  Visco soft contact lens: Viso soft contact lens or one of the study lenses on two eyes and follow up for 3 months (90 days). It is necessary to remove contact lenses every day and replace after 30 days.
- Biofinity Soft Contact Lens: Comfilcon A, Daily wear, monthly disposable soft contact lens
  Biofinity soft contact lens: Biofinity soft contact lens or one of the study lenses on two eyes and follow up for 3 months (90 days). It is necessary to remove contact lenses every day and replace after 30 days.
Period: Overall Study
Arm/Group | Visco Soft Contact Lens | Biofinity Soft Contact Lens
Started | 40 | 20
Completed | 40 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Visco Soft Contact Lens | Biofinity Soft Contact Lens | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 20 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.15 (6.44) | 36.30 (5.53) | 34.87 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 17 | 52
  Male | 5 | 3 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 40 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Visual acuity correctable to snellen 20/25 or better
Time Frame: 3 months
Measure: Count of Units; unit: eye
Units Other Than Participants: eye
Arm/Group | Visco Soft Contact Lens | Biofinity Soft Contact Lens
Number analyzed (Participants) | 40 | 20
Number analyzed (eye) | 80 | 40
eye | 80 | 40

2. Secondary Outcome: Slit Lamp Findings
Description: Any slit lamp finding > Grade 2; Measured on a scale of 0-4 with 0=no findings and 4=severe findings
Time Frame: 3 month
Measure: Count of Units; unit: eye
Units Other Than Participants: eye
Arm/Group | Visco Soft Contact Lens | Biofinity Soft Contact Lens
Number analyzed (Participants) | 40 | 20
Number analyzed (eye) | 80 | 40
eye | 0 | 0

3. Secondary Outcome: Symptoms, Problems and Complaints and Incidence Rate
Description: Subjective Responses to comfort/symptoms/complaints were measured at every visit. 1=Severe Burning to 10=No Burning for each eye
Time Frame: 3 month
Measure: Count of Units; unit: eye
Units Other Than Participants: eye
Arm/Group | Visco Soft Contact Lens | Biofinity Soft Contact Lens
Number analyzed (Participants) | 40 | 20
Number analyzed (eye) | 80 | 40
eye | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Visco Soft Contact Lens | Biofinity Soft Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 0/40 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No